CLINICAL TRIAL: NCT07053865
Title: Electromyographic Assessment of Sleep Bruxism in Patients With Stage III and IV Periodontitis: Findings From a Cross-sectional Study.
Brief Title: Electromyographic Assessment of Sleep Bruxism in Patients With Stage III and IV Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Nicola Discepoli, Associate Professor, University of Siena
Other Study IDs: PB001
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Bruxism; Periodontitis; Sleep Bruxism
MeSH Terms: conditions — Bruxism; Periodontitis; Sleep Bruxism | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontitis Group: Patients diagnosed with Stage III or IV periodontitis according to the 2017 World Workshop classification. Participants will undergo full-mouth periodontal examination and 24-hour surface EMG recording of the masseter muscle to assess sleep bruxism activity.
  Interventions: Device: Surface Electromyography (dia-BRUXO)
- Healthy Control Group: Participants without clinical signs of periodontal disease, matched by age and sex to the periodontitis group. They will also receive a full-mouth periodontal screening and 24-hour surface EMG recording of the masseter muscle for sleep bruxism assessment.
  Interventions: Device: Surface Electromyography (dia-BRUXO)

INTERVENTIONS:
Device: Surface Electromyography (dia-BRUXO) — Participants will undergo 24-hour surface electromyographic recording of the left masseter muscle using the dia-BRUXO portable device to quantify sleep bruxism activity through Bruxism Work Index (BWI) and Bruxism Time Index (BTI).

SUMMARY:
This study aims to investigate the association between periodontitis Stage III and IV and the intensity and duration of sleep bruxism episodes. Surface electromyography (EMG) of the masseter muscle will be used to instrumentally assess sleep bruxism in patients with and without periodontal disease

DETAILED DESCRIPTION:
The purpose of this cross-sectional study is to evaluate whether patients with Stage III and IV periodontitis exhibit differences in sleep bruxism activity compared to individuals without periodontal disease. Participants will undergo comprehensive periodontal assessment and 24-hour EMG recording of the masseter muscle using a portable device. Bruxism activity will be quantified using the Bruxism Work Index (BWI) and Bruxism Time Index (BTI). The study aims to clarify the potential relationship between periodontal inflammation and masticatory muscle activity during sleep, following standardized diagnostic and recording protocols

ELIGIBILITY:
Inclusion Criteria:

* Age between 28 and 50 years
* Ability to perform adequate oral hygiene
* Willingness to participate and sign informed consent
* For periodontitis group: Diagnosis of Stage III or IV periodontitis
* For control group: Absence of periodontal disease

Exclusion Criteria:

* Use of removable dentures
* Ongoing orthodontic treatment
* Temporomandibular disorders (TMD) or orofacial pain
* Use of medications affecting muscle activity
* Systemic or psychiatric disorders
* Diabetes

Ages: 28 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients and healthy controls aged 28-50 years recruited at the University of Siena, Italy. The study includes both individuals with advanced periodontitis and healthy controls.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Sleep Bruxism Work Index (BWI) | Within 24 hours after EMG device application
  BWI is calculated as the percentage of muscle work exerted during bruxism-related masticatory activity relative to the theoretical maximum work. It will be used to assess the intensity of sleep bruxism based on EMG recordings of the masseter muscle

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Discepoli, DDS, PhD, Principal Investigator — Department of Medical Biotechnologies, University of Siena
Locations (1):
- AOUS, Siena, Italy